CLINICAL TRIAL: NCT07131618
Title: The Effect of Cryocompression on Peripheral Neuropathy in Patients Receiving Chemotherapy for Gynecological Cancer
Acronym: CryoPN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, burcu okayer özer, MSc, PhD(c), Registered Nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/302
Record Dates: First submitted 2025-08-05; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Gynecological Cancers; Peripheral Neuropathy Due to Chemotherapy
Keywords: Gynecological cancer; cryocompression; peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental)
  Interventions: Other: cryocompression
- control (No Intervention)

INTERVENTIONS:
Other: cryocompression — Cryocompression induces vasoconstriction in the applied area, thereby reducing blood flow. As a result, the delivery of the chemotherapeutic agent to peripheral nerves is limited, and it is aimed to protect nerve tissue from toxic effects. At the same time, low temperature slows down nerve conduction and cellular metabolism, helping to prevent damage to nerve cells.
  30 minutes after the start of the paclitaxel infusion, cryocompression will be applied using ice gel gloves for the hands and socks for the feet, lasting 30 minutes. After paclitaxel ends, carboplatin will be infused intravenously in 250 cc isotonic solution over 1 hour. Cryocompression will again be applied 30 minutes after the start of the carboplatin infusion using the same method, for 30 minutes. This intervention will be performed weekly during each cycle of the 6-week carboplatin/paclitaxel protocol, for a total of 60 minutes per session.
  Arms: intervention

SUMMARY:
Study Design:

This study is designed as a prospective, randomized controlled experimental study aiming to determine the effect of cryocompression therapy, applied during chemotherapy, on peripheral neuropathy symptoms in women with gynecologic cancers.

Research Hypotheses:

* H₀: Cryocompression therapy has no effect on peripheral neuropathy.
* H₁: Cryocompression therapy has an effect on peripheral neuropathy.

Study Population:

The study population will consist of women over the age of 18 living in Mersin, Türkiye, who are diagnosed with gynecologic cancer and undergoing chemotherapy between August 10 and December 31, 2025.

DETAILED DESCRIPTION:
This study will be conducted with women diagnosed with gynecological cancer who apply to the Oncology Outpatient Clinic and Ambulatory Chemotherapy Unit of Mersin University Hospital and voluntarily agree to participate in the research.

The sample size was calculated using the G*Power 3.1.9.7 program, based on the Chi-Square Test of Independence. In a previous study, the incidence of peripheral neuropathy was reported as 28.2% in the cold therapy group and 57.5% in the control group. Using these data, with a 5% margin of error (α = 0.05) and 80% power (1-β = 0.80), the required sample size was determined to be 35 participants per group. Considering potential data loss, the sample size in each group was increased by approximately 10%, resulting in 39 participants per group. A total of 78 participants will be included in the study.

Inclusion Criteria:

Age 18 years or older,

Diagnosed with gynecological cancer,

Receiving weekly carboplatin-paclitaxel chemotherapy protocol,

Willing to participate in the study and signing the informed consent form.

Intervention:

Participants will be randomly assigned into two groups:

Intervention Group: Cryocompression will be applied during chemotherapy using glove- and sock-shaped cryotherapy devices. The application will begin 15 minutes before the start of chemotherapy infusion, continue during chemotherapy administration, and last for an additional 15 minutes after infusion completion.

Control Group: Standard chemotherapy treatment will be administered without any additional intervention.

Data Collection Process:

After obtaining ethics committee approval, eligible women who meet the study criteria and agree to participate will be given verbal and written information about the study. The informed consent form will be included on the first page of the data collection tool. Those who sign the consent form will complete the questionnaire, which is expected to take approximately 10 minutes.

Study Timeline:

Participant recruitment will begin on August 10, 2025, and will be completed by December 31, 2025.

ELIGIBILITY:
Inclusion Criteria:

* Applying to Mersin University Hospital Oncology Outpatient Clinic
* Willing to participate and providing signed informed consent
* Able to read and write in Turkish
* Accessible and able to communicate
* Citizen of the Republic of Türkiye
* Diagnosed with gynecologic cancer (ovarian, endometrial, or cervical) and aged ≥18 years
* Receiving weekly carboplatin + paclitaxel chemotherapy protocol
* No subjective peripheral neuropathy symptoms before starting chemotherapy
* No history of peripheral neuropathy related to previous taxane/platinum-based chemotherapy protocols
* No psychiatric disorders
* No diseases that may cause peripheral neuropathy such as diabetes, rheumatoid arthritis, or fibromyalgia

Exclusion Criteria:

* Not applying to the specified outpatient clinic
* No gynecologic cancer diagnosis or younger than 18 years old
* Not providing informed consent
* Not receiving weekly carboplatin + paclitaxel chemotherapy protocol
* Presence of subjective peripheral neuropathy symptoms before starting chemotherapy
* History of peripheral neuropathy related to previous taxane/platinum-based chemotherapy protocols
* Presence of psychiatric disorders
* Having diseases that may cause peripheral neuropathy such as diabetes, rheumatoid arthritis, or fibromyalgia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 78 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-Induced Peripheral Neuropathy Assessment Tool | One week after each chemotherapy cycle (6 weeks total).
  Change in peripheral neuropathy severity measured by the Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) Scale range: 0 to 80 (higher scores indicate more severe neuropathy symptoms). Time Frame: One week after each weekly chemotherapy cycle, for six cycles (total 6 weeks).
  Description: Peripheral neuropathy severity will be assessed using the CIPNAT scale, which evaluates sensory, motor, and autonomic symptoms associated with chemotherapy-induced peripheral neuropathy. Scores from all six cycles will be summed for analysis.

IPD SHARING:
Plan to Share IPD: Yes
IPD Sharing Description: Individual participant data (IPD) will not be shared publicly. However, de-identified data may be shared with qualified researchers upon reasonable request, provided that appropriate ethical approvals are obtained.
  IPD Sharing Time Frame: Upon request, after the publication of the main results.
  IPD Sharing Access Criteria: Requests will be evaluated on a case-by-case basis and will be subject to institutional and ethics committee approval.
  IPD Sharing Supporting Information: The study protocol and statistical analysis plan may also be shared.
Supporting Information: Study Protocol
Time Frame: The IPD will be available within 6 months after publication of the primary results and will remain accessible for up to 5 years.
Access Criteria: Access will be granted to qualified researchers affiliated with academic or clinical institutions upon submission of a research proposal, signing of a data use agreement, and approval by the principal investigator and relevant ethics committee.

REFERENCES:
- [Background] Molnar M, Rigo J Jr, Hertelendy F. Signal transduction in human myometrial cells. Acta Physiol Hung. 1996;84(2):89-97. PMID 9046355
- [Background] Scotte F, Tourani JM, Banu E, Peyromaure M, Levy E, Marsan S, Magherini E, Fabre-Guillevin E, Andrieu JM, Oudard S. Multicenter study of a frozen glove to prevent docetaxel-induced onycholysis and cutaneous toxicity of the hand. J Clin Oncol. 2005 Jul 1;23(19):4424-9. doi: 10.1200/JCO.2005.15.651. PMID 15994152
- [Background] Paprocka M, Budzynski W, Kusnierczyk H, Radzikowski C. Effect of cyclophosphamide on mouse bone marrow and leukemic stem cells. Arch Immunol Ther Exp (Warsz). 1980;28(3):447-51. PMID 7447649
- [Background] Hoki T. [The significance of limbal reaction for corneal antigen-antibody reaction]. Nihon Ganka Kiyo. 1966 Jul;17(7):721-31. No abstract available. Japanese. PMID 6007752